CLINICAL TRIAL: NCT07236632
Title: Hyaluronic Acid Versus Botox Injection in Treatment of Life Long Drug Resistant Premature Ejaculation. Which is Better? Randomized Study
Brief Title: Hyaluronic Acid vs Botulinum Toxin Injection in Treatment of Lifelong Drug-Resistant Premature Ejaculation: Randomized Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Maher Wahba, Assistant Lecturer of Urology, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD 9-5-2025
Record Dates: First submitted 2025-11-15; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Premature Ejaculation
Keywords: Hyaluronic Acid; Botulinum Toxins; Ejaculation; Glans Penis; Bulbospongiosus Muscle; Intradermal Injections; Drug Resistance
MeSH Terms: conditions — Premature Ejaculation | interventions — Botulinum Toxins, Type A; Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: Two-arm randomized trial comparing botulinum toxin A injection into the bulbospongiosus muscle vs hyaluronic acid injection into the glans (Fanning Technique) in lifelong drug-resistant premature ejaculation (PE).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinum Toxin Injection Group (Experimental): Participants in this group will receive intramuscular injection of botulinum toxin type A into the bulbospongiosus muscle. A total dose of 100 units of botulinum toxin type A, diluted in 10 milliliters of normal saline, will be administered under ultrasound guidance. The injection will be divided equally, with 5 milliliters injected on each side of the muscle to ensure even distribution across most muscle fibers. The procedure will be performed under aseptic conditions with patients in the lithotomy position.
  Interventions: Drug: Botulinum toxin type A
- Hyaluronic Acid Injection Group (Experimental): Participants in this group will receive injection of hyaluronic acid into the glans penis using the Fanning Technique. Two milliliters of 3.5 percent micronized hyaluronic acid gel will be injected through a single puncture site using a 27-gauge needle. The injection will start from the tip of the glans and proceed toward the coronal sulcus to achieve uniform distribution of the gel. The procedure will be performed under local anesthesia with application of topical lidocaine and prilocaine cream for 30 minutes prior to injection.
  Interventions: Drug: Hyaluronic acid

INTERVENTIONS:
Drug: Botulinum toxin type A — Botulinum toxin type A will be reconstituted by diluting 100 units in 10 milliliters of sterile normal saline. Using ultrasound guidance, 5 milliliters will be injected into each side of the bulbospongiosus muscle through a single puncture site while the patient is in the lithotomy position. The aim is to achieve even distribution of the toxin within the muscle fibers to reduce muscular contractions associated with ejaculation.
  Arms: Botulinum Toxin Injection Group
Drug: Hyaluronic acid — Two milliliters of 3.5 percent micronized hyaluronic acid gel will be injected into the dermis of the glans penis using the Fanning Technique. The injection will be performed through a single puncture site with a 27-gauge needle, advancing from the tip of the glans toward the coronal sulcus to distribute the gel evenly. Topical anesthetic cream containing lidocaine and prilocaine will be applied for 30 minutes before the procedure.
  Arms: Hyaluronic Acid Injection Group

SUMMARY:
Premature ejaculation (PE) is one of the most common male sexual dysfunctions, often resistant to conventional pharmacological and behavioral treatments. This randomized clinical trial aims to compare the safety and efficacy of two minimally invasive treatment options - hyaluronic acid (HA) injection into the glans penis versus botulinum toxin type A injection into the bulbospongiosus muscle - in men with lifelong drug-resistant premature ejaculation. Eighty participants will be randomly assigned in a 1:1 ratio to receive either HA or botulinum toxin injection. The primary outcome is change in intravaginal ejaculatory latency time (IELT). Secondary outcomes include changes in Premature Ejaculation Diagnostic Tool (PEDT), Arabic Index of Premature Ejaculation (AIPE) scores, Premature Ejaculation Profile (PEP), patient satisfaction, and treatment-related adverse events during a 12-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Adult male patients aged 22 to 45 years.
* Sexually active and in a stable heterosexual relationship.
* Circumcised.
* Able to understand and comply with study procedures and follow-up visits.
* Diagnosed with lifelong drug-resistant premature ejaculation, defined as persistent ejaculation within one minute of penetration despite prior pharmacologic or behavioral therapy.
* Normal serum total testosterone, prolactin, and thyroid-stimulating hormone levels.
* Willing to provide written informed consent.

Exclusion Criteria:

* Presence or history of erectile dysfunction or other sexual or ejaculatory disorders such as retrograde ejaculation or acquired premature ejaculation.
* History of acute or chronic prostatitis.
* Any debilitating medical condition including hepatic failure, renal failure, or uncontrolled diabetes mellitus.
* Previous pelvic or spinal surgery.
* Prior chemotherapy or radiotherapy.
* Use of antipsychotic or neuroactive medications that may affect ejaculation.
* History of substance abuse or current drug dependence.
* Presence of penile prosthesis, penile deformity, or anatomic abnormalities of the glans or shaft.
* Known hypersensitivity or allergy to botulinum toxin or hyaluronic acid preparations.
* Any condition that, in the investigator's opinion, may interfere with the safety or evaluation of the study treatment.

Ages: 22 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in intravaginal ejaculatory latency time | Baseline, 1 month, 3 months, 6 months, and 12 months after intervention
  The duration from vaginal penetration to ejaculation will be recorded using a stopwatch by the patient's partner. The median intravaginal ejaculatory latency time will be calculated for each participant from several intercourse attempts. The change in latency time after treatment compared with baseline will be used to assess treatment efficacy.

SECONDARY OUTCOMES:
Change in Premature Ejaculation Diagnostic Tool (PEDT) score | Baseline, 1 month, 3 months, 6 months, and 12 months after intervention
  The Premature Ejaculation Diagnostic Tool questionnaire will be used to evaluate changes in ejaculatory control and distress levels. Higher scores indicate greater severity.
Change in Arabic Index of Premature Ejaculation (AIPE) score | Baseline, 1 month, 3 months, 6 months, and 12 months after intervention
  The Arabic Index of Premature Ejaculation questionnaire will assess subjective improvement in control, satisfaction, and distress related to ejaculation. Higher scores reflect better control and lower distress.
Change in Premature Ejaculation Profile (PEP) score | Baseline, 1 month, 3 months, 6 months, and 12 months after intervention
  The Premature Ejaculation Profile will be used to evaluate treatment-related improvement across four domains: perceived control, personal distress, interpersonal difficulty, and sexual satisfaction.
Patient satisfaction score | 1 month, 3 months, 6 months, and 12 months after intervention
  Participants will rate overall satisfaction with the procedure using a four-point scale (0 = dissatisfied, 1 = slightly satisfied, 2 = satisfied, 3 = very satisfied).

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in this study will be made available to qualified researchers upon reasonable request. Shared data will include demographic characteristics, intervention details, and outcome measures related to intravaginal ejaculatory latency time, questionnaire scores, and adverse events. No information that could identify participants will be released.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified data will be available beginning six months after publication of the primary results and will remain accessible for up to three years.
Access Criteria: Researchers may submit a formal request to the principal investigator describing the intended analyses and data use. Requests will be reviewed by the study steering committee. Data will be shared electronically in compliance with institutional and ethical guidelines.